CLINICAL TRIAL: NCT06125509
Title: Defining Intervention Targets Along Pathways From Cumulative Stress and Trauma to Alcohol and HIV Self-management Among Young People Living With HIV (Project DEFINE)
Brief Title: SHARE Project Define
Status: Completed | Type: Observational
Sponsor: Florida State University (Other)
Collaborators: University of California, San Diego (Other); Nova Southeastern University (Other); University of Florida (Other); University of Central Florida (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sylvie Naar, Principal Investigator, Florida State University
Other Study IDs: STUDY00002535; 1P01AA029547-01 (NIH)
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of the current study is to define modifiable intervention targets that are developmentally- and culturally-relevant in pathways between cumulative stress and self-management outcomes - alcohol use and HIV - among Young People Living with HIV (YPLWH).

This is a correlational, longitudinal cohort study that will seek to evaluate the association of cumulative stress with self-management of alcohol (i.e. hazardous drinking) and HIV (viral suppression) among YPLWH. The study will enroll up to 175 participants between the ages of 18-29 who currently reside in Florida and are living with HIV.

In the Model phase, individuals will participate in two assessment timepoints, including baseline assessment with a two-week sleep diary completion and 9-month follow-up assessment with another two-week sleep diary completion. The aim of the model phase is to define key modifiable intervention targets by longitudinally evaluating multiple components of sleep health, and emotion and behavioral regulation among YPLWH to determine potential pathways between cumulative stress and alcohol and HIV outcomes, in the context of individual factors relevant to YPLWH (e.g., age, race/ethnicity, cannabis and other substance use, cognitive functioning, education), with an additional cross-project moderator aim to explore age, biological sex and gender, race/ethnicity, other substance use, and mental health as moderators.

In the Adapt phase, 42 of N=175 will participate in 60-90 minute focus groups, that will focus on adapting developmentally and culturally scalable measures of cumulative stress, sleep health, and emotion/behavior regulation for screening and intervention targeting, and creation of a community-informed toolkit of the adapted measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and 0 months to 29 years and 11 months
* Currently reside in Florida
* Report having had at least 1 alcoholic drink in the last 30 days
* Able to read and understand English
* Have internet access via smartphone, tablet or computer
* Be diagnosed as HIV positive and;
* Willing to provide informed consent.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults
* Individuals who are not diagnosed as HIV+
* Prisoners
* Pregnant women

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adults aged 18-29 who reside in Florida and are living with HIV and report having had at least 1 alcoholic drink in the last 30 days (see inclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Alcohol Use | 9 months
  Hazardous Drinking
HIV Viral Load | 9 months
  Viral Suppression

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Center for Translational Behavioral Science, Tallahassee, Florida, United States